CLINICAL TRIAL: NCT07247981
Title: T1 Tissue Mapping as a Non Invasive Biomarker for Quantification of Chronic Thyroid Related Microscopic Myocardial Fibrosis.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lina Mohamed Farid, Lina Mohamed Farid, Assiut University
Other Study IDs: CMR T1 tissue mapping
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Thyroid Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CMR T1 tissue mapping helps in detection and quantification of the microscopic myocardial fibrosis and is more accurate and non invasive maneuver.

DETAILED DESCRIPTION:
Chronic thyroid diseased patients either hypo or hyperthyroidism may develop arrhythmias or even atrial fibrillation which is worrisome. And since early detection provides the early management, T1 tissue mapping of the heart provides accurate quantification of the myocardial fibrosis throughout the imaged organ.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic thyroid disease.

Exclusion Criteria:

* patients with other chronic illnesses ( diabetes, hypertension, .. etc).
* patients received neck radiation therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hypo and hyperthyroidism in both genders.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial fibrosis | 1 year
  Detection and quantification of myocardial fibrosis.